CLINICAL TRIAL: NCT00886522
Title: Intrabone Infusion of Cord Blood Hemopoietic Stem Cells in Adult Patients With High Risk Haematological Malignancies.
Brief Title: Intrabone Infusion of Cord Blood in Adults With Hematological Malignancies
Acronym: IBCB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Francesca Bonifazi, MD, MD, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 152/2008/U/Sper
Record Dates: First submitted 2009-04-22; First posted 2009-04-23 (Estimated); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Hematological Malignancies
Keywords: Anti-thymocyte globulin Fresenius; Busulfan; Cord blood; Cyclophosphamide; Fludarabine; Human Leucocyte Antigen; Hematopoietic Stem Cell; Hematopoietic Stem Cell Transplant; Graft-versus-Host-Disease; Graft-versus-Host-Disease prophylaxis; Intrabone infusion; Thiotepa
MeSH Terms: conditions — Hematologic Neoplasms; Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intrabone cord blood infusion (Experimental): All adults patients with hematological malignancies, lacking a HLA matched donor but with a HLA compatible CB unit, fulfilling the inclusion criteria, will undergo to intrabone HSC infusion of CB.
  Interventions: Procedure: Intrabone cord blood infusion

INTERVENTIONS:
Procedure: Intrabone cord blood infusion — Myeloablative conditioning regimen (MAC):
  i.v. Busulfan 12.8 mg/kg, Cyclophosphamide 120 mg/kg, ATG-Fresenius 30 mg/kg
  Reduced intensity conditioning regimen (RIC):
  Tiothepa 10 mg/kg, Fludarabine 100 mg/kg, Cyclophosphamide 100 mg/kg, ATG-Fresenius 30 mg/kg
  GVHD prophylaxis:
  Cyclosporine 1 mg/kg since day -7 to +120, Mycophenolate 15 mg kg x 2 since day +1 to +27

SUMMARY:
The purpose of this study is to evaluate the engraftment of donor hemopoiesis (proportion of transplanted patients with successful engraftment at day +42) in adult patients affected by high risk hematological malignancies after intrabone infusion of cord blood.

DETAILED DESCRIPTION:
For many hematological malignancies, hemopoietic stem cell (HSC) transplant is the only possible treatment. The source of HSC is often bone marrow (BM) or, in the past 10 years, peripheral blood cell (PBSC) mobilized by granulocyte growth factor. Transplant needs a HLA compatible (related or unrelated) donor. Around 10-30% of patients with indication for allogeneic HSC transplant are not able to undergo the procedure because of the lack of a HLA compatible donor. Cord blood (CB) cells represent another possible source, which needs a lower degree of HLA compatibility, this type of transplant, however, offers a lower number of HSC. For this reason, adult patients, until now, could not use this source, because of the not suitable number of cell per kg, of recipient body weight. Recently, in experimental animal models it was observed that intrabone HSC transplant allows, in the recipient, engraftment of donor hemopoiesis by using a 1Log (10-1) lower number of cells compared to the intravenous way (Yahata 2003, Castello 2004). Safety and feasibility of intrabone infusion was verified by two clinical studies on humans: the first was conducted by Ringden O. et al. in 18 patients without any evidence of collateral effects and with complete engraftment of donor hemopoiesis with BM as a source of HSC (Hagglund 1998); the second one was conducted by Frassoni et al. (Frassoni 2008) with CB as the source of HSC.

The aim of this study is to evaluate the intrabone infusion instead of the intravenous one, for the HSC transplant from CB in patients with haematological malignancies when it is not possible to find a HLA matched donor.

We will perform:

* evaluation of the engraftment kinetics;
* evaluation of the chimerism degree at 30, 60, 100 days, 6 months and 1 year after transplant;
* studies on immunological reconstitution and the role of the NK compartment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years.
* Patients affected by hematological malignancies without a HLA identical sibling donor or unrelated donor.
* Informed consent.

Exclusion Criteria:

* Patients with ECOG < 2.
* Patients with blood creatine > 2 mg/dl or with transaminase or cholestase index > 5 times compared to normality upper limits.
* Patients with Cardiac Fraction Ejection < 40%.
* Patients with DLCO < 60% or Diffusing Lung Capacity of carbon monoxide attesting a severe pulmonary insufficiency.
* Patients with peripheral blast cell count over 10%.
* Second neoplasia diagnosed no more than 2 years before.
* Patients with active or suspected infection by fungi for which a therapeutic treatment is ongoing.
* HIV positive patients.
* HCV-RNA and HBV-RNA positive patients (it is possible to enrol them after discussion with the Principal Investigator).
* Pregnant or lactating women.
* Severe mental diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-04; Primary Completion 2012-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Proportion of transplanted patients with successful engraftment at day +42 | Within the first 42 days

SECONDARY OUTCOMES:
Clinical response with the analysis of global survival, survival without relapse, relapse incidence | 1 year
Acute and chronic GVHD incidence | For acute GVHD 100 days; for chronic GVHD 1 year
Infection incidence | 1 year
Chimerism study on selected populations (myeloid, lymphoid, NK) | 30, 60, 100 days, 6 months and 1 year
Studies on immunological reconstitution | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Bonifazi, MD, Principal Investigator — S. Orsola-Malpighi University Hospital
Locations (1):
- Hematology Institute "L. and A. Seràgnoli", S. Orsola-Malpighi University Hospital, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ballen KK, Spitzer TR, Yeap BY, McAfee S, Dey BR, Attar E, Haspel R, Kao G, Liney D, Alyea E, Lee S, Cutler C, Ho V, Soiffer R, Antin JH. Double unrelated reduced-intensity umbilical cord blood transplantation in adults. Biol Blood Marrow Transplant. 2007 Jan;13(1):82-9. doi: 10.1016/j.bbmt.2006.08.041. PMID 17222756
- [Background] Barker JN, Davies SM, DeFor T, Ramsay NK, Weisdorf DJ, Wagner JE. Survival after transplantation of unrelated donor umbilical cord blood is comparable to that of human leukocyte antigen-matched unrelated donor bone marrow: results of a matched-pair analysis. Blood. 2001 May 15;97(10):2957-61. doi: 10.1182/blood.v97.10.2957. PMID 11342417
- [Background] Barker JN, Weisdorf DJ, DeFor TE, Blazar BR, Miller JS, Wagner JE. Rapid and complete donor chimerism in adult recipients of unrelated donor umbilical cord blood transplantation after reduced-intensity conditioning. Blood. 2003 Sep 1;102(5):1915-9. doi: 10.1182/blood-2002-11-3337. Epub 2003 May 8. PMID 12738676
- [Background] Barker JN, Weisdorf DJ, DeFor TE, Blazar BR, McGlave PB, Miller JS, Verfaillie CM, Wagner JE. Transplantation of 2 partially HLA-matched umbilical cord blood units to enhance engraftment in adults with hematologic malignancy. Blood. 2005 Feb 1;105(3):1343-7. doi: 10.1182/blood-2004-07-2717. Epub 2004 Oct 5. PMID 15466923
- [Background] Bradley MB, Satwani P, Baldinger L, Morris E, van de Ven C, Del Toro G, Garvin J, George D, Bhatia M, Roman E, Baxter-Lowe LA, Schwartz J, Qualter E, Hawks R, Wolownik K, Foley S, Militano O, Leclere J, Cheung YK, Cairo MS. Reduced intensity allogeneic umbilical cord blood transplantation in children and adolescent recipients with malignant and non-malignant diseases. Bone Marrow Transplant. 2007 Oct;40(7):621-31. doi: 10.1038/sj.bmt.1705785. Epub 2007 Jul 30. PMID 17660841
- [Background] Brunstein CG, Barker JN, Weisdorf DJ, DeFor TE, Miller JS, Blazar BR, McGlave PB, Wagner JE. Umbilical cord blood transplantation after nonmyeloablative conditioning: impact on transplantation outcomes in 110 adults with hematologic disease. Blood. 2007 Oct 15;110(8):3064-70. doi: 10.1182/blood-2007-04-067215. Epub 2007 Jun 14. PMID 17569820
- [Background] Cornetta K, Laughlin M, Carter S, Wall D, Weinthal J, Delaney C, Wagner J, Sweetman R, McCarthy P, Chao N. Umbilical cord blood transplantation in adults: results of the prospective Cord Blood Transplantation (COBLT). Biol Blood Marrow Transplant. 2005 Feb;11(2):149-60. doi: 10.1016/j.bbmt.2004.11.020. PMID 15682076
- [Background] Cohen Y, Nagler A. Umbilical cord blood transplantation--how, when and for whom? Blood Rev. 2004 Sep;18(3):167-79. doi: 10.1016/S0268-960X(03)00064-X. PMID 15183901
- [Background] De Witte T, Van Biezen A, Hermans J, Labopin M, Runde V, Or R, Meloni G, Mauri SB, Carella A, Apperley J, Gratwohl A, Laporte JP. Autologous bone marrow transplantation for patients with myelodysplastic syndrome (MDS) or acute myeloid leukemia following MDS. Chronic and Acute Leukemia Working Parties of the European Group for Blood and Marrow Transplantation. Blood. 1997 Nov 15;90(10):3853-7. PMID 9354651
- [Background] Dick JE and Lapidot T. Stem cells take a shortcut to the bone marrow. Blood 2003(101):2901-2902.
- [Background] Eapen M, Rubinstein P, Zhang MJ, Stevens C, Kurtzberg J, Scaradavou A, Loberiza FR, Champlin RE, Klein JP, Horowitz MM, Wagner JE. Outcomes of transplantation of unrelated donor umbilical cord blood and bone marrow in children with acute leukaemia: a comparison study. Lancet. 2007 Jun 9;369(9577):1947-54. doi: 10.1016/S0140-6736(07)60915-5. PMID 17560447
- [Background] Fanning LR, Hegerfeldt Y, Tary-Lehmann M, Lesniewski M, Maciejewski J, Weitzel RP, Kozik M, Finney M, Lazarus HM, Paul P, Ratajczak MZ, Meyerson HJ, Laughlin MJ. Allogeneic transplantation of multiple umbilical cord blood units in adults: role of pretransplant-mixed lymphocyte reaction to predict host-vs-graft rejection. Leukemia. 2008 Sep;22(9):1786-90. doi: 10.1038/leu.2008.55. Epub 2008 Mar 20. No abstract available. PMID 18354493
- [Background] Frassoni F, Gualandi F, Podestà M et al. Direct intra-bone injection of unrelated cord blood cells overcomes the problem of delayed/failure to engraft and improves the feasibility of haematopoietic transplant in adult patients. Bone Marrow Transp 41(81):21, 2008.
- [Background] Gluckman E, Broxmeyer HA, Auerbach AD, Friedman HS, Douglas GW, Devergie A, Esperou H, Thierry D, Socie G, Lehn P, et al. Hematopoietic reconstitution in a patient with Fanconi's anemia by means of umbilical-cord blood from an HLA-identical sibling. N Engl J Med. 1989 Oct 26;321(17):1174-8. doi: 10.1056/NEJM198910263211707. No abstract available. PMID 2571931
- [Background] Gluckman E, Rocha V, Arcese W, Michel G, Sanz G, Chan KW, Takahashi TA, Ortega J, Filipovich A, Locatelli F, Asano S, Fagioli F, Vowels M, Sirvent A, Laporte JP, Tiedemann K, Amadori S, Abecassis M, Bordigoni P, Diez B, Shaw PJ, Vora A, Caniglia M, Garnier F, Ionescu I, Garcia J, Koegler G, Rebulla P, Chevret S; Eurocord Group. Factors associated with outcomes of unrelated cord blood transplant: guidelines for donor choice. Exp Hematol. 2004 Apr;32(4):397-407. doi: 10.1016/j.exphem.2004.01.002. PMID 15050751
- [Background] Gluckman E, Rocha V, Boyer-Chammard A, Locatelli F, Arcese W, Pasquini R, Ortega J, Souillet G, Ferreira E, Laporte JP, Fernandez M, Chastang C. Outcome of cord-blood transplantation from related and unrelated donors. Eurocord Transplant Group and the European Blood and Marrow Transplantation Group. N Engl J Med. 1997 Aug 7;337(6):373-81. doi: 10.1056/NEJM199708073370602. PMID 9241126
- [Background] Goldstone AH, Burnett AK, Wheatley K, Smith AG, Hutchinson RM, Clark RE; Medical Research Council Adult Leukemia Working Party. Attempts to improve treatment outcomes in acute myeloid leukemia (AML) in older patients: the results of the United Kingdom Medical Research Council AML11 trial. Blood. 2001 Sep 1;98(5):1302-11. doi: 10.1182/blood.v98.5.1302. PMID 11520775
- [Background] Greenberg P, Cox C, LeBeau MM, Fenaux P, Morel P, Sanz G, Sanz M, Vallespi T, Hamblin T, Oscier D, Ohyashiki K, Toyama K, Aul C, Mufti G, Bennett J. International scoring system for evaluating prognosis in myelodysplastic syndromes. Blood. 1997 Mar 15;89(6):2079-88. PMID 9058730
- [Background] Grewal SS, Barker JN, Davies SM, Wagner JE. Unrelated donor hematopoietic cell transplantation: marrow or umbilical cord blood? Blood. 2003 Jun 1;101(11):4233-44. doi: 10.1182/blood-2002-08-2510. Epub 2003 Jan 9. No abstract available. PMID 12522002
- [Background] Hagglund H, Ringden O, Agren B, Wennberg L, Remberger M, Rundquist L, Svahn BM, Aspelin P. Intraosseous compared to intravenous infusion of allogeneic bone marrow. Bone Marrow Transplant. 1998 Feb;21(4):331-5. doi: 10.1038/sj.bmt.1701116. PMID 9509965
- [Background] Hansen JA and Dupont B. HLA 2004 Immunobiology of the Human MHC. Proceedings of the 13th IHWC. IHWG Press 2004, Seattle, WA (USA).
- [Background] Horwitz ME, Morris A, Gasparetto C, Sullivan K, Long G, Chute J, Rizzieri D, McPherson J, Chao N. Myeloablative intravenous busulfan/fludarabine conditioning does not facilitate reliable engraftment of dual umbilical cord blood grafts in adult recipients. Biol Blood Marrow Transplant. 2008 May;14(5):591-4. doi: 10.1016/j.bbmt.2008.02.016. PMID 18410902
- [Background] Josefson A. A new method of treatment - intraossal injections. Acta Med Scand 1934; 81:550-564.
- [Background] Komatsu T, Narimatsu H, Yoshimi A, Kurita N, Kusakabe M, Hori A, Murashige N, Matsumura T, Kobayashi K, Yuji K, Tanaka Y, Kami M. Successful engraftment of mismatched unrelated cord blood transplantation following reduced intensity preparative regimen using fludarabine and busulfan. Ann Hematol. 2007 Jan;86(1):49-54. doi: 10.1007/s00277-006-0190-5. Epub 2006 Oct 12. PMID 17036221
- [Background] Kurtzberg J, Laughlin M, Graham ML, Smith C, Olson JF, Halperin EC, Ciocci G, Carrier C, Stevens CE, Rubinstein P. Placental blood as a source of hematopoietic stem cells for transplantation into unrelated recipients. N Engl J Med. 1996 Jul 18;335(3):157-66. doi: 10.1056/NEJM199607183350303. PMID 8657213
- [Background] Laughlin MJ, Barker J, Bambach B, Koc ON, Rizzieri DA, Wagner JE, Gerson SL, Lazarus HM, Cairo M, Stevens CE, Rubinstein P, Kurtzberg J. Hematopoietic engraftment and survival in adult recipients of umbilical-cord blood from unrelated donors. N Engl J Med. 2001 Jun 14;344(24):1815-22. doi: 10.1056/NEJM200106143442402. PMID 11407342
- [Background] List AF, Vardiman J, Issa JP, DeWitte TM. Myelodysplastic syndromes. Hematology Am Soc Hematol Educ Program. 2004:297-317. doi: 10.1182/asheducation-2004.1.297. PMID 15561689
- [Background] Locatelli F, Giorgiani G, Giraldi E, Castelnovi C, Stroppa P, Bernardo ME, Bonetti F, Maccario R. Cord blood transplantation in childhood. Haematologica. 2000 Nov;85(11 Suppl):26-9. No abstract available. PMID 11268320
- [Background] Long GD, Laughlin M, Madan B, Kurtzberg J, Gasparetto C, Morris A, Rizzieri D, Smith C, Vredenburgh J, Halperin EC, Broadwater G, Niedzwiecki D, Chao NJ. Unrelated umbilical cord blood transplantation in adult patients. Biol Blood Marrow Transplant. 2003 Dec;9(12):772-80. doi: 10.1016/j.bbmt.2003.08.007. PMID 14677117
- [Background] Lowenberg B, Suciu S, Archimbaud E, Haak H, Stryckmans P, de Cataldo R, Dekker AW, Berneman ZN, Thyss A, van der Lelie J, Sonneveld P, Visani G, Fillet G, Hayat M, Hagemeijer A, Solbu G, Zittoun R. Mitoxantrone versus daunorubicin in induction-consolidation chemotherapy--the value of low-dose cytarabine for maintenance of remission, and an assessment of prognostic factors in acute myeloid leukemia in the elderly: final report. European Organization for the Research and Treatment of Cancer and the Dutch-Belgian Hemato-Oncology Cooperative Hovon Group. J Clin Oncol. 1998 Mar;16(3):872-81. doi: 10.1200/JCO.1998.16.3.872. PMID 9508168
- [Background] Mazurier F, Doedens M, Gan OI, Dick JE. Rapid myeloerythroid repopulation after intrafemoral transplantation of NOD-SCID mice reveals a new class of human stem cells. Nat Med. 2003 Jul;9(7):959-63. doi: 10.1038/nm886. PMID 12796774
- [Background] Mayer RJ, Davis RB, Schiffer CA, Berg DT, Powell BL, Schulman P, Omura GA, Moore JO, McIntyre OR, Frei E 3rd. Intensive postremission chemotherapy in adults with acute myeloid leukemia. Cancer and Leukemia Group B. N Engl J Med. 1994 Oct 6;331(14):896-903. doi: 10.1056/NEJM199410063311402. PMID 8078551
- [Background] Migliaccio AR, Adamson JW, Stevens CE, Dobrila NL, Carrier CM, Rubinstein P. Cell dose and speed of engraftment in placental/umbilical cord blood transplantation: graft progenitor cell content is a better predictor than nucleated cell quantity. Blood. 2000 Oct 15;96(8):2717-22. PMID 11023503
- [Background] Moretta A, Maccario R, Fagioli F, Giraldi E, Busca A, Montagna D, Miniero R, Comoli P, Giorgiani G, Zecca M, Pagani S, Locatelli F. Analysis of immune reconstitution in children undergoing cord blood transplantation. Exp Hematol. 2001 Mar;29(3):371-9. doi: 10.1016/s0301-472x(00)00667-6. PMID 11274766
- [Background] Mori T, Aisa Y, Nakazato T, Yamazaki R, Shimizu T, Mihara A, Yamane A, Ikeda Y, Okamoto S. Tacrolimus and methotrexate for the prophylaxis of graft-versus-host disease after unrelated donor cord blood transplantation for adult patients with hematologic malignancies. Transplant Proc. 2007 Jun;39(5):1615-9. doi: 10.1016/j.transproceed.2006.12.042. PMID 17580201
- [Background] Narimatsu H, Kami M, Miyakoshi S, Murashige N, Yuji K, Hamaki T, Masuoka K, Kusumi E, Kishi Y, Matsumura T, Wake A, Morinaga S, Kanda Y, Taniguchi S. Graft failure following reduced-intensity cord blood transplantation for adult patients. Br J Haematol. 2006 Jan;132(1):36-41. doi: 10.1111/j.1365-2141.2005.05832.x. PMID 16371018
- [Background] Narimatsu H, Terakura S, Matsuo K, Oba T, Uchida T, Iida H, Hamaguchi M, Watanabe M, Kohno A, Murata M, Sawa M, Miyamura K, Morishita Y. Short-term methotrexate could reduce early immune reactions and improve outcomes in umbilical cord blood transplantation for adults. Bone Marrow Transplant. 2007 Jan;39(1):31-9. doi: 10.1038/sj.bmt.1705539. Epub 2006 Nov 20. PMID 17115066
- [Background] Narimatsu H, Watanabe M, Kohno A, Sugimoto K, Kuwatsuka Y, Uchida T, Murata M, Miyamura K, Morishita Y; Nagoya Blood and Marrow Transplantation Group (NBMTG). High incidence of graft failure in unrelated cord blood transplantation using a reduced-intensity preparative regimen consisting of fludarabine and melphalan. Bone Marrow Transplant. 2008 Apr;41(8):753-6. doi: 10.1038/sj.bmt.1705978. Epub 2008 Jan 14. No abstract available. PMID 18195683
- [Background] Ooi J, Iseki T, Takahashi S, Tomonari A, Takasugi K, Shimohakamada Y, Yamada T, Ishii K, Ohno N, Nagamura F, Uchimaru K, Tojo A, Asano S. Unrelated cord blood transplantation for adult patients with de novo acute myeloid leukemia. Blood. 2004 Jan 15;103(2):489-91. doi: 10.1182/blood-2003-07-2420. Epub 2003 Aug 21. PMID 12933570
- [Background] Ooi J, Iseki T, Takahashi S, Tomonari A, Ishii K, Takasugi K, Shimohakamada Y, Ohno N, Uchimaru K, Nagamura F, Tojo A, Asano S. Unrelated cord blood transplantation for adult patients with advanced myelodysplastic syndrome. Blood. 2003 Jun 15;101(12):4711-3. doi: 10.1182/blood-2002-12-3917. Epub 2003 Feb 13. PMID 12586621
- [Background] Rocha V, Cornish J, Sievers EL, Filipovich A, Locatelli F, Peters C, Remberger M, Michel G, Arcese W, Dallorso S, Tiedemann K, Busca A, Chan KW, Kato S, Ortega J, Vowels M, Zander A, Souillet G, Oakill A, Woolfrey A, Pay AL, Green A, Garnier F, Ionescu I, Wernet P, Sirchia G, Rubinstein P, Chevret S, Gluckman E. Comparison of outcomes of unrelated bone marrow and umbilical cord blood transplants in children with acute leukemia. Blood. 2001 May 15;97(10):2962-71. doi: 10.1182/blood.v97.10.2962. PMID 11342418
- [Background] Rocha V, Locatelli F. Searching for alternative hematopoietic stem cell donors for pediatric patients. Bone Marrow Transplant. 2008 Jan;41(2):207-14. doi: 10.1038/sj.bmt.1705963. Epub 2007 Dec 17. PMID 18084331
- [Background] Rocha V, Wagner JE Jr, Sobocinski KA, Klein JP, Zhang MJ, Horowitz MM, Gluckman E. Graft-versus-host disease in children who have received a cord-blood or bone marrow transplant from an HLA-identical sibling. Eurocord and International Bone Marrow Transplant Registry Working Committee on Alternative Donor and Stem Cell Sources. N Engl J Med. 2000 Jun 22;342(25):1846-54. doi: 10.1056/NEJM200006223422501. PMID 10861319
- [Background] Rubinstein P, Carrier C, Carpenter C et al. Graft selection in unrelated placental/umbilical cord blood (PCB) transplantation: influence and weight of HLA match and cell dose on engraftment and survival [abstract]. Blood 2000; 96:588a.
- [Background] Rubinstein P, Stevens CE. Placental blood for bone marrow replacement: the New York Blood Center's program and clinical results. Baillieres Best Pract Res Clin Haematol. 2000 Dec;13(4):565-84. doi: 10.1053/beha.2000.0106. PMID 11102277
- [Background] Talvensaari K, Clave E, Douay C, Rabian C, Garderet L, Busson M, Garnier F, Douek D, Gluckman E, Charron D, Toubert A. A broad T-cell repertoire diversity and an efficient thymic function indicate a favorable long-term immune reconstitution after cord blood stem cell transplantation. Blood. 2002 Feb 15;99(4):1458-64. doi: 10.1182/blood.v99.4.1458. PMID 11830500
- [Background] Uchida N, Wake A, Takagi S, Yamamoto H, Kato D, Matsuhashi Y, Matsumura T, Seo S, Matsuno N, Masuoka K, Kusumi E, Yuji K, Miyakoshi S, Matsuzaki M, Yoneyama A, Taniguchi S. Umbilical cord blood transplantation after reduced-intensity conditioning for elderly patients with hematologic diseases. Biol Blood Marrow Transplant. 2008 May;14(5):583-90. doi: 10.1016/j.bbmt.2008.03.003. PMID 18410901
- [Background] van Hennik PB, de Koning AE, Ploemacher RE. Seeding efficiency of primitive human hematopoietic cells in nonobese diabetic/severe combined immune deficiency mice: implications for stem cell frequency assessment. Blood. 1999 Nov 1;94(9):3055-61. PMID 10556189
- [Background] Wagner JE, Barker JN, DeFor TE, Baker KS, Blazar BR, Eide C, Goldman A, Kersey J, Krivit W, MacMillan ML, Orchard PJ, Peters C, Weisdorf DJ, Ramsay NK, Davies SM. Transplantation of unrelated donor umbilical cord blood in 102 patients with malignant and nonmalignant diseases: influence of CD34 cell dose and HLA disparity on treatment-related mortality and survival. Blood. 2002 Sep 1;100(5):1611-8. doi: 10.1182/blood-2002-01-0294. PMID 12176879
- [Background] Wattel E, Solary E, Leleu X, Dreyfus F, Brion A, Jouet JP, Hoang-Ngoc L, Maloisel F, Guerci A, Rochant H, Gratecos N, Casassus P, Janvier M, Brice P, Lepelley P, Fenaux P. A prospective study of autologous bone marrow or peripheral blood stem cell transplantation after intensive chemotherapy in myelodysplastic syndromes. Groupe Francais des Myelodysplasies. Group Ouest-Est d'etude des Leucemies aigues myeloides. Leukemia. 1999 Apr;13(4):524-9. doi: 10.1038/sj.leu.2401387. PMID 10214857
- [Background] Yahata T, Ando K, Sato T, Miyatake H, Nakamura Y, Muguruma Y, Kato S, Hotta T. A highly sensitive strategy for SCID-repopulating cell assay by direct injection of primitive human hematopoietic cells into NOD/SCID mice bone marrow. Blood. 2003 Apr 15;101(8):2905-13. doi: 10.1182/blood-2002-07-1995. Epub 2002 Oct 31. PMID 12411299
- [Derived] Bonifazi F, Dan E, Labopin M, Sessa M, Guadagnuolo V, Ferioli M, Rizzi S, De Carolis S, Sinigaglia B, Motta MR, Bontadini A, Giudice V, Martinelli G, Arpinati M, Cavo M, Bonafe M, Storci G. Intrabone transplant provides full stemness of cord blood stem cells with fast hematopoietic recovery and low GVHD rate: results from a prospective study. Bone Marrow Transplant. 2019 May;54(5):717-725. doi: 10.1038/s41409-018-0335-x. Epub 2018 Sep 19. PMID 30232415
- See also: The European Group for Blood and Marrow Transplantation — http://www.ebmt.org/
- See also: Italian Group for Bone Marrow Transplantation and Cellular Therapy — http://www.gitmo.net/